CLINICAL TRIAL: NCT02782546
Title: A Phase II Study of Cytokine Induced Memory-like NK Cell Adoptive Therapy After Haploidentical Donor Hematopoietic Cell Transplantation
Brief Title: Cytokine Induced Memory-like NK Cell Adoptive Therapy After Haploidentical Donor Hematopoietic Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); The V Foundation for Cancer Research (Other); National Cancer Institute (NCI) (NIH); ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201610088; 1P50CA171963-01A1 (NIH); 2P50CA171963-06 (NIH)
Record Dates: First submitted 2016-05-22; First posted 2016-05-25 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Tacrolimus; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; ALT-803; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recipient (Experimental): * Standard of care reduced conditioning regimen on Day -1
  * Graft cell infusion on Day 0
  * Post-transplant cyclophosphamide on Days +3 and +4
  * GvHD prophylaxis with tacrolimus and mycophenolate mofetil (MMF) will start on Day +5. MMF will continue till Day +35 and tacrolimus till Day +180 in the absence of GvHD
  * G-CSF will start on Day +7 and will continue until neutrophil engraftment as per institutional guidelines
  * The cytokine-induced memory like natural killer (CIML NK) cells will be infused on Day +7 without a filter or pump, slowly by gravity over at least 15 minutes.
  * ALT-803 will start approximately 4 hours after the CIML NK cell infusion. ALT-803 will be administered subcutaneously at a dose of 10 mcg/kg subcutaneously beginning Day +7 (on the day of CIML NK cell infusion) and then every 21 days for a total of 4 doses
  Interventions: Procedure: Graft cell infusion; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: G-CSF; Procedure: CIML NK cell infusion; Drug: ALT-803
- Donor (Experimental): * Donors will receive subcutaneous G-CSF from Day -4 till Day 0 and undergo 20L apheresis per institutional guidelines.
  * Two consecutive days for collection are allowed in case of the target CD34+ cell dose being less than the target 4 x106/kg-bw from the first day of collection.
  * On Day +6 (one day before the planned CIML NK cell infusion), peripheral blood mononuclear cells will be collected by a single standard 20-L apheresis over 4-5 hours from the same haploidentical related donor that provided the HCT graft.
  Interventions: Procedure: Leukapheresis

INTERVENTIONS:
Procedure: Graft cell infusion — -Day 0
  Other Names: HCT
  Arms: Recipient
Drug: Tacrolimus — -GVHD prophylaxis
  Other Names: Prograf
  Arms: Recipient
Drug: Mycophenolate mofetil — -GVHD prophylaxis
  Other Names: CellCept; Myfortic
  Arms: Recipient
Drug: G-CSF — -Continue until neutrophil engraftment as per institutional guidelines
  Other Names: Granulocyte-colony stimulating factor
  Arms: Recipient
Procedure: CIML NK cell infusion — -Day +7
  Arms: Recipient
Drug: ALT-803 — -Start approximately 4 hours after CIML NK cell infusion
  Arms: Recipient
Procedure: Leukapheresis — -Day +6
  Arms: Donor

SUMMARY:
This is a standard phase 2 study powered to demonstrate improvement in the 100 day leukemia free survival to 30% from <10% expected with the use of reduced intensity haplo-HCT in this extremely high-risk patient cohort (based on the institutional experience using non-myeloablative / reduced intensity conditioning in a similar patient cohort).

A formal safety evaluation will be done after every 6th patient enrolled and the trial will be stopped if noted to have unusually higher engraftment failure (acute GVHD rates (>60% any grades or >30% grade III/IV or ≥ 50% severe cGVHD) or engraftment failure rates (≥15%).

ELIGIBILITY:
Recipient Inclusion Criteria:

* Refractory AML without complete remission (CR) after 2 or more cycles of induction therapy (primary induction failure), or AML relapsed after obtaining a CR and failed one or more cycles of re-induction therapy. Standard dose 10-day decitabine (20 mg/m2 daily IV x 10 days) or 7-day azacitidine (75-100 mg/m2 daily SC/IV x 7 days) will be considered as one cycle of induction therapy.
* At least 18 years of age
* Available HLA-haploidentical donor that meets the criteria in the protocol
* Patients with known CNS involvement with AML are eligible provided that they have been treated and CSF is clear for at least 2 weeks prior to enrollment into the study. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.
* Karnofsky performance status > 60 %
* Adequate organ function as defined below:

  * Total bilirubin < 2 mg/dl
  * AST(SGOT)/ALT(SGPT) < 3.0 x IULN
  * Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m2 by Cockcroft-Gault Formula
  * Oxygen saturation ≥90% on room air and adjusted DLCO of at least 40%
  * Ejection fraction ≥40%
* Able to be off of corticosteroids (10 mg or less of prednisone or equivalent doses of other systemic steroids are allowed) and any other immune suppressive medications beginning on Day -3
* Women of childbearing potential must have a negative pregnancy test within 28 days prior to study registration. Female and male patients (along with their female partners) must agree to use two forms of acceptable contraception, including one barrier method, during participation in the study and throughout the DLT evaluation period.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Recipient Exclusion Criteria:

* Relapsed after allogeneic transplantation.
* Circulating blast count >30,000/uL by morphology or flow cytometry (cyto-reductive therapies including leukapheresis or hydroxyurea are allowed).
* Uncontrolled bacterial or viral infections, or known HIV, Hepatitis B or C infection.
* Presence of donor specific antibodies (DSA) with Mean Fluorescence Intensity (MFI) of >5000 as assessed by the single antigen bead assay, < 6 weeks prior to starting transplant conditioning
* Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
* New progressive pulmonary infiltrates on screening chest x-ray or chest CT scan that have not been evaluated with bronchoscopy. Infiltrates attributed to infection must be stable/ improving after 1 week of appropriate therapy (4 weeks for presumed or proven fungal infections)
* Known hypersensitivity to one or more of the study agents
* Received any investigational drugs within the 14 days prior to the first day of transplant conditioning
* Pregnant and/or breastfeeding

Donor Inclusion Criteria:

* Related donor (sibling, offspring, or offspring of sibling)
* At least 18 years of age
* HLA-haploidentical donor/recipient match by at least Class I serologic typing at the A&B locus.
* In general good health, and medically able to tolerate leukapheresis required for harvesting the NK cells for this study.
* Ability to understand and willingness to sign an IRB approved written informed consent document

Donor Exclusion Criteria:

* Positive for hepatitis, HTLV, or HIV infection
* Pregnant and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2028-02-13 (Estimated)

PRIMARY OUTCOMES:
Leukemia free survival rate (LFS) | 1 year post transplantation
  -LFS is defined as the time from achievement of CR to the time of relapse, death in remission, or last follow-up.

SECONDARY OUTCOMES:
Leukemia free survival rate (LFS) | 3 months post transplantation
  -LFS is defined as the time from achievement of CR to the time of relapse, death in remission, or last follow-up.
Rate of overall survival (OS) | 1 year post transplantation
  -OS is defined as the time from the date of Day 0 until death from any cause.
Incidence of relapse in patients who are found to be CR (complete remission) | Day 28 post transplantation
  -CR: Morphologically leukemia free state (i.e. bone marrow with <5% blasts by morphologic criteria and no blasts with Auer rods, no evidence of extramedullary leukemia) and absolute neutrophil count ≥1000 /μL and platelets ≥100,000 /μL. Patient must be independent of transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berrien-Elliott MM, Foltz JA, Russler-Germain DA, Neal CC, Tran J, Gang M, Wong P, Fisk B, Cubitt CC, Marin ND, Zhou AY, Jacobs MT, Foster M, Schappe T, McClain E, Kersting-Schadek S, Desai S, Pence P, Becker-Hapak M, Eisele J, Mosior M, Marsala L, Griffith OL, Griffith M, Khan SM, Spencer DH, DiPersio JF, Romee R, Uy GL, Abboud CN, Ghobadi A, Westervelt P, Stockerl-Goldstein K, Schroeder MA, Wan F, Lie WR, Soon-Shiong P, Petti AA, Cashen AF, Fehniger TA. Hematopoietic cell transplantation donor-derived memory-like NK cells functionally persist after transfer into patients with leukemia. Sci Transl Med. 2022 Feb 23;14(633):eabm1375. doi: 10.1126/scitranslmed.abm1375. Epub 2022 Feb 23. PMID 35196021
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu